CLINICAL TRIAL: NCT05800873
Title: A Phase 1b/2 Study To Evaluate The Efficacy, Safety, Pharmacokinetics And Pharmacodynamics Of EVER001 In Participants With Selected Proteinuric Glomerular Diseases
Brief Title: Evaluate The Efficacy, Safety, Pharmacokinetics And Pharmacodynamics Of EVER001
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Everest Medicines (China) Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ES108001
Record Dates: First submitted 2023-03-09; First posted 2023-04-06 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Primary Membranous Nephropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EVER001 100mg (Experimental): EVER001 100mg QD for 4 weeks, followed by EVER001 100mg BID for 32 weeks.
  Interventions: Drug: EVER001
- EVER001 200mg (Experimental): EVER001 200mg BID for 36 weeks.
  Interventions: Drug: EVER001

INTERVENTIONS:
Drug: EVER001 — A highly selective, oral, reversable, covalent Bruton tyrosine kinase (BTK) inhibitor with high selectivity over other kinases.
  Arms: EVER001 100mg
Drug: EVER001 — A highly selective, oral, reversable, covalent Bruton tyrosine kinase (BTK) inhibitor with high selectivity over other kinases.
  Arms: EVER001 200mg

SUMMARY:
EVER001 is a highly selective, oral, reversable, covalent Bruton tyrosine kinase (BTK) inhibitor with high selectivity over other kinases, which is being developed to treat proteinuric glomerular diseases.

The overall aim of the study is to evaluate the efficacy, safety, pharmacokinetics and pharmacodynamics of EVER001 in subjects with selected proteinuric glomerular diseases. The first targeted disease is primary membranous nephropathy.

ELIGIBILITY:
Inclusion Criteria:

1. Having clinical diagnosis of primary membranous nephropathy, as verified by biopsy.
2. Have positive anti-PLA2R autoantibody test results > 20 relative units (RU)/ml.
3. During screening at least one testing of proteinuria must be >3.5 g/24h.
4. Have nephrotic range proteinuria for at least 8 weeks prior to Day 1 and no improvement (<50% reduction) despite supportive therapy of ACE inhibitor or ARB unless contraindicated, for patients who have two tests of proteinuria during screening ≥8.0g/24h, the duration of nephrotic range proteinuria for at least 8 weeks is not required.

Exclusion Criteria:

1. Non-primary membranous nephropathy or other condition affecting the kidney.
2. eGFR at screening < 45 mL/min/1.73m2 or kidney function not stable .
3. Uncontrolled hypertension .
4. Serum albumin level at screening # 25g/l.
5. Have received: B-cell targeted therapy except rituximab at any time;Rituximab and the biosimilars within 2 years (participants with rituximab treatment between 1 and 2 years prior to Day 1 are eligible if there is documented evidence of B-cell repopulation to >90% of Lower Limits of Normal Range.); Cyclophosphamide or Chlorambucil within 180 days;other immunosuppressive/immunomodulatory agents within 90 days;greater than 30mg/day prednisone or equivalence within 30 days.
6. Acute or chronic infection,including positivity of tuberculosis infection test.
7. Positive serology for TP,HIV, HBV, or HCV.
8. Lab testing abnormality as: WBC< 3000/mm³, Lymphocyte < 1000/ mm³, neutrophil <1500/mm³, Hb < 80g/L, Platelet count <100×10e9/ L, Prothrombin time>1.5×ULN, Activated partial thromboplastin time ≥1.5×ULN, Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≥ 1.5×ULN, alkaline phosphatase and bilirubin >1.5×ULN.
9. Judged by the investigator that the participant is unlikely to comply with study procedures, restrictions, and requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
adverse events | 104 weeks.
clinical laboratory assessments. | 104 weeks.
vital signs. | 104 weeks.
physical examination | 104 weeks
ECG. | 104 weeks.

SECONDARY OUTCOMES:
To evaluate whether EVER001 can modulate proteinuria in pMN. | 52 weeks.
  Percentage change from baseline of 24 hr proteinuria throughout 52 weeks.
To evaluate whether EVER001 can modulate anti-PLA2R autoantibodies in patients with positive baseline levels of these antibodies. | 52 weeks.
  Percentage change from baseline of anti-PLA2R autoantibody level throughout 52 weeks.
To evaluate the clinical response and immunological response in pMN. | 104 weeks.
  To evaluate the clinical response and immunological response in pMN.
Maximum Observed Plasma Concentration (Cmax) of EVER001 | 52 weeks.
Minimum Observed Plasma Concentration (Cmin) of EVER001 | 52 weeks.
Time to Reach Maximum Observed Concentration (Tmax) of EVER001. | 52 weeks.

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - The Second Xiangya Hospital Of Central South University, Changsha, Changsha
  - The First Affiliated Hospital of PLA Army Medical University, Chongqing, Chongqing Municipality
  - The Third Affiliated Hospital,Sun Yat Sen University, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Harbin
  - Xiangya Third Hospital, Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Medical college of Xi'an Jiaotong University, Xian, Shanxi
  - Sichuan Province People's Hospital, Chengdu, Sichuan
  - Second Hospital of Shanxi Medical University, Shanxi, Taiyuan
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - The first affliated hospital of NingBo university, Ningbo, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - Peking University First Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No